CLINICAL TRIAL: NCT04092686
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled, Fixed-dose, Multicenter Study to Evaluate the Efficacy and Safety of SEP-363856 in Acutely Psychotic Subjects With Schizophrenia
Brief Title: A Clinical Trial That Will Study the Efficacy and Safety of an Investigational Drug in Acutely Psychotic People With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 361-302; 2019-000697-37 (EudraCT Number)
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: acute psychosis; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, parallel-group, placebo-controlled, fixed-dose, multicenter study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEP-363856 75mg (Experimental): SEP-363856 75mg dosed once daily
  Interventions: Drug: SEP-363856 75mg
- SEP-363856 100mg (Experimental): SEP-363856 100mg dosed once daily
  Interventions: Drug: SEP-363856 100mg
- Placebo (Placebo Comparator): Placebo dosed once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-363856 75mg — SEP-363856 75mg tablet dosed once daily
  Arms: SEP-363856 75mg
Drug: SEP-363856 100mg — SEP-363856 100mg tablet dosed once daily
  Arms: SEP-363856 100mg
Drug: Placebo — Placebo tablet dosed once daily
  Arms: Placebo

SUMMARY:
A clinical trial to study the efficacy and safety of an investigational drug in acutely psychotic people with schizophrenia. Participants in the study will either receive the drug being studied or a placebo. This study is accepting male and female participants between 18 -65 years old who have been diagnosed with schizophrenia. This study will be conducted in 60 locations world wide. The study will last up to nine (9) weeks.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group, fixed-dosed study evaluating the efficacy and safety of two doses of SEP-363856 (75 and 100 mg/day) versus placebo over a 6-week Treatment Period in acutely psychotic subjects with schizophrenia. This study is projected to randomize approximately 462 subjects to 3 treatment groups (SEP-363856 75 mg/day, SEP-363856 100 mg/day, or placebo) in a 1:1:1 ratio. Treatment assignment will be stratified by country. Study drug will be taken once a day and may be taken with or without food.

This study is designed to test the hypotheses that treatment with SEP-363856 in adult subjects with schizophrenia will result in significantly greater reduction (i.e. improvement) in PANSS total score and CGI-S score at Week 6 from Baseline when compared to placebo. The overall Type I error is controlled for two hierarchical families of hypotheses. The first family includes hypotheses about the testing of change from Baseline in PANSS total score at Week 6 between each of the SEP-363856 dose levels vs. placebo. The second family of hypotheses are about the testing of change from Baseline in CGI-S score at Week 6 between each of the SEP-363856 dose levels vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject between 18 to 65 years of age (inclusive) at the time of consent.
2. Subject must give written informed consent and privacy authorization prior to participation in the study; adolescents must also provide informed assent.
3. Subject meets DSM-5 criteria for schizophrenia as established by clinical interview at screeing.
4. Subject must have a CGI-S score ≥ 4
5. Subject must have a PANSS total score ≥ 80 and a PANSS item score ≥ 4 on 2 or more of the following PANSS items: delusions, conceptual disorganization, hallucinations, and unusual thought content
6. Subject has an acute exacerbation of psychotic symptoms (persisting no longer than 2 months prior to providing informed consent).
7. Subject has marked deterioration of functioning in one or more areas.
8. Subject is, in the opinion of the Investigator, generally healthy based on screening medical history, PE, neurological examination, vital signs, ECG and clinical laboratory values.

Exclusion Criteria:

1. Subject has a DSM-5 diagnosis or presence of symptoms consistent with a DSM-5 diagnosis other than schizophrenia. Exclusionary disorders include but are not limited to alcohol use disorder (within past 12 months), substance (other than nicotine or caffeine) use disorder within past 12 months, or lifetime history of significant substance abuse that, in the opinion of the Investigator or Sponsor, may have had a significant and potentially permanent impact on the brain or other body systems, major depressive disorder, bipolar I or II disorder, schizoaffective disorder, obsessive compulsive disorder, and posttraumatic stress disorder. Symptoms of mild to moderate mood dysphoria or anxiety are allowed so long as these symptoms are not the primary focus of treatment.
2. Subject is at significant risk of harming self, others, or objects based on Investigator's judgment.
3. Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study
4. Female subject who is pregnant or lactating
5. Subject has any clinically significant abnormal laboratory value(s) at Screening as determined by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Positive and negative syndrome scale (PANSS) total score at Endpoint (Week 6) | Baseline and Week 6
  PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210.

SECONDARY OUTCOMES:
Change from Baseline in Clinical Global Impressions - Severity (CGI-S) score at Endpoint (Week 6) | Baseline and Week 6
  The CGI-S is a single-item clinician-rated assessment of the subject's current illness state on a 7-point scale (score range: 1-7), where a higher score is associated with greater illness severity.

CONTACTS AND LOCATIONS:
Locations (62):
- United States (18):
  - Woodland Research Northwest, Rogers, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - Clinical Innovations, Inc., Bellflower, California
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, Long Beach, California
  - California Neuropsychopharmacology Clinical Research Institute, San Diego, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Larkin Behavioral Health Services, Hollywood, Florida
  - South Florida Research Phase I-IV, INC., Miami Springs, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Pillar Clinical Research, Chicago, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - CBH Health, LLC, Gaithersburg, Maryland
  - Arch Clinical Trials, LLC, St Louis, Missouri
  - Hassman Research Institute, Marlton, New Jersey
  - New York State Psychiatric Institute, New York, New York
  - Pillar Clinical Research, Richardson, Texas
- Bulgaria (6):
  - Mental Health Centre, Prof. Dr. Ivan Temkov, Burgas EOOD, Department for Treatment of Emergency Psychiatric Conditions, Burgas
  - State Psychiatric Hospital - Kardzhali, First Woman Department, Third Men Deparment, Kardzhali
  - State Psychiatric Hospital Sv. Ivan rilski-Department General Psychiatry for Adults "closed" Type -Men, Department General Psychiatry for Adults, "Closed" Type - Women, Novi Iskar
  - UMHAT Sveti Georgi EAD, Plovdiv
  - Mental Health Center - Sofia EOOD Unit for Active Treatment of Persons with Serious Mental Disorders, Sofia
  - UMHAT Alexandrovska EAD Second Department of Pshychiatry at Clinic of Psychiatry, Sofia
- Psychiatric Hospital "Sveti Ivan", Zagreb, Croatia
- Latvia (3):
  - LTD Psychoeurological Hospital of Daugavpils, Daugavpils
  - SLLC Riga Centre of Psychiatry and Narcology, Riga
  - SLLC Psychoneurological Hospital of Strenci, Strenči
- Russia (13):
  - State Budgetary Healthcare Institution of Arkhangelsk region "Arkhangelsk clinical psychiatric hospital", Arkhangelsk
  - State Healthcare Institution "Psychiatric Hospital of Engels" of MoH of Saratov Region, departments № 1 and 3, 166, Engel's
  - State Budgetary Institution of Healthcare of Moscow "Psychiatric Clinical Hospital #1 named after N.A. Alekseev of Department of Healthcare of Moscow, Moscow
  - State Budgetary Institution of Healthcare of Moscow "Psychiatric Hospital No. 5", Moscow
  - State Public Institution of Healthcare Leningrad Regional Psychoneurological Dispensary, Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare "Psychiatric Hospital named after P.P. Kashchenko, inpatient No 2 leg add, Saint Petersburg
  - FSBI "NMRC of Psychiatry and Neurology named after V.M. Bekterev" MoH RF, Saint Petersburg
  - FSBI- "NMRC of Psychiatry and Neurology named after V.M. Bekhterev" MoH RF3, Saint Petersburg
  - Saint Petersburg State Public Institution of Healthcare "City Psychiatric Hospital #3 named after I.I. Skvortsov-Stepanov", Saint Petersburg
  - State Institution of Healthcare "Saratov City Clinical Hospital #2 named after V.I. Razumovskiy" 20 and 21 departments, Saratov
  - State Institution of Healthcare Regional Clinical Psychiatric Hospital of Saint Sofia, Saratov
  - State Budgetary Healthcare Institution of Stavropol region "Stavropol Region Psychiatric Hospital # 2", Stavropol
  - Federal State Budgetary Scientific Institution "Tomsk National Research Medical Center of Russian Academy of Sciences",, Tomsk
- Serbia (11):
  - Clinic of Psychiatry, Clinical Center of Serbia,, Belgrade
  - Clinic of Psychiatry, Clinical Center of Serbia, Belgrade
  - Clinical Center "Dr Dragisa Misovic- Dedinje", Belgrade
  - Special Hospital for Psychiatric Diseases "Kovin", Kovin
  - Special Neuropsychiatric Hospital Kovin, Kovin
  - Clinic of Psychiatry, clinical Center Kragujevac, Kragujevac
  - University Clinical Center Kragujevac, Clinic of Psychiatry, Kragujevac
  - University Clinical Center Nis, Clinic of Psychiatry, Niš
  - Special Hospital for Psychiatric Disease Sveti Vracevi, Novi Kneževac
  - Special Hospital for Psychiatric Diseases "SVeti Vracevi", Novi Kneževac
  - Special Hospital for Psychiatric Diseases "Dr Slavoljub Bakalovic", Vršac
- Ukraine (10):
  - 46 Academician Pavlov St, Kharkiv
  - State Institution Institute of Neurology, Psychiatry and Narcology of the National Academy of Medical Sciences of Ukraine, Department of Boundary Psychiatry, Kharkiv
  - Communica Noncommercial Enterprise Kherson Regional Institution of Psychiatric Care Assistance of Kherson Regional Council, Male Department of Psychiatry #3, Female Department of Psychiatry #10, Kherson
  - Kyev Clinical Hospital on Railway Station #1 of Healthcare Center branch of JSC "Ukrainian railway" Department of Psychoneurology, Kyiv
  - National Military and Medical Clinical Center, The Main Military Clinical Hospital, Psychiatric Clinic with Wards for Narcological Patients, Kyiv
  - Communal Institution of Kyiv Regional Council Regional Psychiatric and Narcological Medical Association, Male Department #10, Female Department #2, Kyiv
  - Communal Non-commercial Enterprise Kyiv City Psychoneurological Hospital #3 of Executive Body of Kyiv City Council (Kyiv City State Administration), General Psychiatric Department #4 ,, Kyiv
  - Communal Non-commercial Enterprise Kyiv City Psychoneurological Hospital #3 of Executive Body of Kyiv City Council (Kyiv City State Administration), General Psychiatric Department #4, Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Concil Lviv Regional Clinical Psychiatric Hospital, Department #20, Lviv
  - Communal Institution O.I. Yuschenko Vinnytsia Regional Psychoneurological Hospital, Male Department #21, Female Department #15, M.I. Pyrogov Vinnytsia National Medical University, Chair of Psychiatry, Narcology and Psychotherapy with Postgraduate Educatio, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com